CLINICAL TRIAL: NCT05817474
Title: Efficacy of Local Infiltration of Tranexamic Acid and Lidocaine in Tonsillar Bed on Postoperative Bleeding and Pain During Tonsillectomy Surgery.
Brief Title: Efficacy of Local Infiltration of Tranexamic Acid and Lidocaine in Tonsillar Bed on Postoperative Bleeding and Pain During Tonsillectomy Surgery: Prospective, Randomized, Control Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: mohamed (Other)
Collaborators: Al-Azhar University (Other)
Responsible Party: Sponsor-Investigator, mohamed, assissant professor of anesthesia, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mohamed
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Post Operative Pain; Postoperative Hemorrhage
Keywords: Tonsillectomy; Lidocaine
MeSH Terms: conditions — Pain, Postoperative; Postoperative Hemorrhage | interventions — Lidocaine; Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group T (Experimental): Group T: received lidocaine (2 %) 2 ml and tranexamic acid 2 ml in each tonsillar bed;
  Interventions: Drug: lidocaine (2 %) 2 ml and tranexamic acid
- Group N (Placebo Comparator): Group N (Control group): received 4 ml of normal saline in each tonsillar bed.
  Interventions: Drug: lidocaine (2 %) 2 ml and tranexamic acid

INTERVENTIONS:
Drug: lidocaine (2 %) 2 ml and tranexamic acid — lidocaine (2 %) 2 ml and tranexamic acid 2 ml in each tonsillar bed

SUMMARY:
All anesthetic techniques aim to lessen intra-operative surgical site bleeding because it is a major problem and does not help with precision, surgery time, or postoperative wound healing. The main reason for reoperation and mortality in children who have had tonsillectomies is post-tonsillectomy hemorrhage. Pre-emptive analgesia reduces surgical pain blocking of central sensitization by topical or systemic medications.

DETAILED DESCRIPTION:
The control of postoperative pain in children after tonsillectomy is a crucial issue. After a tonsillectomy, it is crucial to receive enough postoperative analgesia since discomfort limits swallowing, increases the risk of dehydration, infection, and subsequent bleeding, and can impede a quick recovery and painless convalescence. Immediately following surgery and during the first 24th hours, this pain is at its most intense (1).

The main reason for reoperation and mortality in children who have had tonsillectomy is post-tonsillectomy hemorrhage (PTH). These two categories of PTH as primary bleeding in the first 24 hours and secondary bleeding (after 24th hours). Most PTH cases are secondary, with incidence reaching its peak between days 5 and 7 after surgery when the fibrin clot breaks from the tonsillar fossa. PTH requiring surgical intervention will be an emergency that most anesthesiologists will encounter in their clinical practice (2).

In numerous surgical procedures, bleeding has been observed to be reduced by antifibrinolytic transexamic acid (3). It has been demonstrated that transexamic acid can reduce blood loss during tonsillectomy but has no impact on whether PTH develops in tonsillectomy patients. When administered by nebulization in the emergency room to a patient who was 3 years old, tranexamic acid has been found to reduce secondary PTH (4).

Plasminogen activation is competitively inhibited by tranexamic acid. As a result of inhibition of the fibrinolysis, it prevents the clots from being broken down thereby significantly reducing surgical hemorrhage. After surgical stress, fibrinolysis occurs more frequently, especially in complex surgeries like total knee arthroplasty. Fibrinolysis reaches its peak six hours after surgery and continues to occur at a high rate for up to 18 hours. When administered during this time, tranexamic acid can significantly less blood loss (5). In those who are predisposed, thrombosis risk from tranexamic acid exists. Orthostatic difficulties, vision abnormalities, headaches, myoclonus, and rash are among other uncommon adverse effects.

The safety and efficacy of tranexamic acid (TXA) have been well studied by surgical services including cardiac, orthopedic, dental, trauma, critical care, and dermatologic surgery. However, except for craniofacial surgery (6). The most serious problems following a tonsillectomy include hemorrhage and respiratory obstruction from edema. The most frequent complaint in the initial post-operative phase is pain. With individual differences, the pain increases anxiety and the fear of swallowing, predisposes to delayed food intake, reduces respiratory effort, increases the risk of pulmonary problems, and lengthens hospital stays (7).

Pre-emptive analgesia, which reduces surgical pain, is the blocking of central sensitization by topical or systemic medications. Opioids, steroids, and NSAIDs have all been tested as pre-emptive analgesics, as well as local anesthetic sprays and infiltration in the tonsillar fossa (8). The use of local anesthetics, opioids, ketamine (9), gabapentin (10), corticosteroids, and even non-pharmacologic interventions as adjuvant local analgesic compounds has been cited frequently in recent years in children undergoing adenotonsillectomy (11).

ELIGIBILITY:
Inclusion criteria

1. Male or female child between 4 and 12 years old
2. ASA one and two, planned for an elective tonsillectomy
3. Patients having 4 or more episodes of tonsillitis in the last year, 5 or more episodes in the previous two years, or 7 episodes in the previous three years.

Exclusion criteria

1-Children with diabetes mellitus, problems of the heart, kidneys, or liver 4-Obstructive sleep apnea syndrome 5-blood disorders, or a propensity to hemorrhage 6-patients suspected of an allergy to the drug being administered, and those undergoing concurrent surgery such as an adenoidectomy or tongue tie.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Postoperative bleeding, pain and postoperative opioid consumption | 12 month
  Postoperative bleeding, pain and postoperative opioid consumption

CONTACTS AND LOCATIONS:
Overall Officials: abdalla mohamed abdalla, MD, Principal Investigator — AZHAR
Locations (1):
- MEDICIN, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided